CLINICAL TRIAL: NCT06120829
Title: Cryobiopsy for Suspected Malignant Peripheral Lymphadenopathy
Acronym: COLD SNAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Goertzen, Pulmonary Critical Care Fellow, San Antonio Uniformed Services Health Education Consortium
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: C.20231002
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cryobiopsy of Peripheral Lymph Nodes
Keywords: Cryobiopsy; Peripheral Lymphadenopathy; Lymphoma; Malignancy Staging
MeSH Terms: conditions — Lymphoma | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (Active Comparator): FNA followed by Core Needle biopsy
  Interventions: Procedure: Core Needle Biopsy
- Experimental Arm (Experimental): FNA followed by cryobiopsy through a introducer sheath
  Interventions: Procedure: Cryobiopsy; Device: Cryobiopsy

INTERVENTIONS:
Procedure: Cryobiopsy — Use of 1.1mm ERBE 2 disposable cryoprobe for tissue sampling
  Arms: Experimental Arm
Device: Cryobiopsy — Use of 1.1mm ERBE 2 disposable cryoprobe for tissue sampling
  Arms: Experimental Arm
Procedure: Core Needle Biopsy — Core Needle Biopsy
  Arms: Control Arm

SUMMARY:
Cryobiopsy of peripheral lymph nodes with suspected malignant potential with comparison to standard core needle biopsy.

DETAILED DESCRIPTION:
Peripheral lymph node biopsy has long been accomplished to establish malignant and non-malignant diagnoses of lymphadenopathy. For several decades patients have undergone fine needle aspiration (FNA) and core needle biopsy (CNB) with patient's proceeding to excisional biopsy if initial less invasive procedures are inadequate. The diagnostic yield of FNA followed by CNB has remained stagnant since the 1990's with a yield range of 66-93.6% depending on multiple factors such as patient factors and malignancy type. In one study they found that between 25-30% of patients undergoing FNA followed by CNB ultimately proceed to excisional biopsy which carries a higher rate of morbidity than FNA or CNB with complications including: Seroma 6.4%, Hematoma 3.2%, Dehiscence 1.8% and prolonged pain 1.4%, vs. CNB which has a less than 1% overall complication rate. In several malignancy types, but especially in lymphoproliferative disorders there is a gap in the ability to diagnose via CNB.

After the introduction of cryobiopsy for bronchoscopic lymph node biopsy there was a significant increase in yields with the most prominent increase seen among the lymphoproliferative disorders with an increase from 69% to 95%. Cryobiopsy samples had a significant increase in architecture which is critical in proper diagnosis of lymphoproliferative disorders and genetic sequencing. Bronchoscopic cryobiopsies of mediastinal lymph nodes did not demonstrate higher complication rates compared to fine needle aspiration despite the higher yields.

Thus far in the literature the use of cryobiopsy for the diagnosis of superficial peripheral lymph nodes of suspected malignant potential has not yet been described. The use of the ERBE 2 platform for tissue biopsy has been demonstrated to improve the diagnostic yield in some situations, such as mediastinal lymphadenopathy, without statistically significant increase in complications. This study seeks to evaluate the safety, feasibility, and effectiveness of the use of the 1.1mm cryoprobe of this platform to increase diagnostic yield of peripherally obtainable lymph nodes of malignant potential without the need for additional procedures such as excisional biopsy that carry a significantly increased risk compared to current initial biopsy methods such as FNA and CNB.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Suspected or confirmed malignancy with suspected involvement of peripheral lymph nodes based on CT, PET-CT or ultrasound imaging with a clinical need for additional tissue or staging by tissue sampling

Exclusion Criteria:

* Age <18 or >89
* Patient preference
* Severe allergy to lidocaine precluding use
* Severe allergy to chlorhexidine precluding use
* Overlying Infection
* Active anticoagulation or anti-platelet therapy, with the exception of aspirin mono-therapy, that cannot be safely held as determined by the performing or prescribing physician.
* Major organs, vasculature or tissue that would preclude the safety of the procedure as determined by the performing physician.
* Inability to reach the lymph node through a core needle introducer sheath as determined by the performing physician.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Yield by strict criteria | 7 days

SECONDARY OUTCOMES:
Complication Rate | 30 days
Patient reported pain on Stanford Comparative Pain Scale | 5 days
Need for Repeat procedures | 30 days
Ability to proceed to next generation sequencing based on tissue obtained | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Following completion of analysis, the electronic medical record query will be destroyed and the Research Database will be de-identified by removing all remaining dates.